CLINICAL TRIAL: NCT04626466
Title: Effect of Irradiation Doses < 10 Gy and of Irradiated Bone Volume on the Variation of Blood Elements of the Complete Blood Count During and After Pelvic Irradiation
Acronym: MIFADORESOL
Status: Completed | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-004; 2020-A01108-31 (Other: IDRCB)
Record Dates: First submitted 2020-11-03; First posted 2020-11-12 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Prostate Carcinoma; Rectum Carcinoma; Anal Canal Carcinoma; Endometrium Carcinoma; Cervix Carcinoma; Radiotherapy; Vaginal Cancer
Keywords: Bone marrow; Hematologic toxicity; Pelvic irradiation; Radiotherapy; Intensity-modulated radiotherapy (IMRT)
MeSH Terms: conditions — Prostatic Neoplasms; Rectal Neoplasms; Anal Canal Carcinoma; Endometrial Neoplasms; Uterine Cervical Neoplasms; Vaginal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-metastatic prostate, rectum, canal, endometrium, cervix or vaginal cancer Radiotherapy treatment
  Interventions: Other: Biological investigations

INTERVENTIONS:
Other: Biological investigations — (complete blood count, platelet count, renal function evaluation)

SUMMARY:
Bone marrow is one of the organs at risk of complications during irradiation due to its radiosensitivity. Hematopoietic toxicity remains one of the main toxicities during irradiation of pelvic lymph node areas, especially when concomitant chemotherapy is used, volume of bone marrow irradiated is large and dose to the bone marrow is high. There is a lack of prospective studies and comparative trials to customize the constraints according to the presence or absence of chemotherapy and correlated to the patient's bone marrow potential. This multicentric and prospective study conducted by Strasbourg Europe Cancerology Institute aims to evaluate hematological toxicity (anemia, thrombocytopenia, leukopenia) in patients treated with pelvic irradiation for prostate, rectum, anal canal, endometrium, cervix cancer or vaginal cancer. One hundred patients will be included in the study, including patients treated with exclusive radiotherapy, radiochemotherapy, or radiohormonal therapy. The primary objective is to quantify the relationship between acute hematological toxicity and delivered doses and irradiated volumes in pelvic bone marrow for pelvic cancers. Hematological toxicity will be measured by weekly blood count during radiotherapy and at one month and three months after the end of radiotherapy. Secondary endpoints are the evaluation of viral, bacterial and fungal infections during and for three months following radiotherapy, as well as the evaluation of the impact of radiation-induced hematological toxicity on the administration of chemotherapy for the concerned patients. The aim of this study is to improve and optimize radiotherapy if a dose limit or volume constraint is imposed by the results of the study.

DETAILED DESCRIPTION:
Patients will be identified as potentially eligible for inclusion once radiotherapy has been decided upon at the multidisciplinary consultation meeting. During the radiotherapy consultation, the study will be offered to the patient if they also meet the other inclusion criteria. As soon as the consent is signed and before the first radiotherapy session, a first biological check-up including a blood count and renal function will be performed. This biological investigation will serve as a reference.

During the dosimetric computer-tomography scan for radiotherapy, bony structures will be delineated, iliac bones, lower pelvis, femoral heads, lumbosacral spine and entire pelvis.

Dosimetry will be performed in the same way whether patients are included in the study or not, they will receive between 25Gy in 5 fractions and 78Gy in 39 fractions, depending on the primary tumor. The dose volume histograms will be received.

During treatment, patients will have a weekly blood test starting from the second week of treatment. At one months and three months after the end of the radiotherapy, patients will be seen in consultation and will also have a blood test.

ELIGIBILITY:
For inclusion in the study, patients must be affiliated to the national or local social security, and must meet all the following criteria :

Inclusion Criteria:

* Patients must be ≥ 18 years old and < 80 years old
* Performance Status 0 to 2
* Histologically-confirmed diagnosis of : prostate cancer ; cervical cancer ; vaginal cancer ; endometrial cancer ; middle or low rectal cancer ; anal duct carcinoma
* At inclusion, patients must have : Haemoglobin > 10 g/dL ; Leucocytes 4.0-11.0 g/L ; Neutrophils 1.5-7.7 g/L ; Platelets 150-400 g/L
* Signed informed consent from the patient

Exclusion Criteria:

* History of haematologic disorders, leucopathia or imune system diseases
* At inclusion, patients must not have : Haemoglobin < 10 g/dL or > 18 g/dL (men) > 16 g/dL (women) ; Leucocytes < 4.0 or > 11.0 g/L ; Neutrophils < 1.5 or > 7.7 g/L ; Platelets < 150 or > 400 g/L
* Patients previously treated with radiation therapy or with chemotherapy
* Patients with metastatic cancer
* Patients presenting tumor classified histologically as sarcomatoid
* Patients placed under judicial protection, guardianship, or supervision
* Women that are pregnant or breast-feeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-metastatic prostate, rectum, anal canal, endometrium, cervix carcinoma or vaginal cancer Radiotherapy treatment validated in a multidisciplinary consultation meeting
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Assessment of acute haematological toxicity according to CTCAE v5.0 | throughout radiotherapy treatment
  * Haemoglobin
  * Platelets
  * Neutrophils
  * Lymphocytes
Assessment of acute haematological toxicity according to CTCAE v5.0 | 1 month after the end of radiotherapy
  * Haemoglobin
  * Platelets
  * Neutrophils
  * Lymphocytes
Assessment of acute haematological toxicity according to CTCAE v5.0 | 3 months after the end of radiotherapy
  * Haemoglobin
  * Platelets
  * Neutrophils
  * Lymphocytes

SECONDARY OUTCOMES:
Number of patients with clinical signs of viral, bacterial, or fungal infections according to CTCAE v5.0 | throughout treatment, at 1 and 3 months
Number of patients undergoing definitive and transient discontinuations of concomitant chemotherapy. | throughout treatment, at 1 and 3 months
Number of patients who required a reduction in chemotherapy dose. | throughout treatment, at 1 and 3 months
Cumulative doses and theoretical doses of chemotherapy. | throughout treatment, at 1 and 3 months
Number of patients undergoing definitive withdrawal or transitory stops of the entire treatment. | throughout treatment, at 1 and 3 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU Jean Minjoz, Besançon
  - Centre Georges François Leclerc, Dijon
  - Institut de Cancerologie Strasbourg Europe, Strasbourg